CLINICAL TRIAL: NCT07166770
Title: Evaluating a Community-Led COVID-19 Testing Intervention to Address Mistrust - Study 2
Brief Title: Community-Led COVID-19 Testing Intervention to Address Mistrust
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Kelli J. England, Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-10-FB-0215 - Study 2
Record Dates: First submitted 2025-09-05; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Trust
Keywords: community-led; COVID-19; trust; vaccine hesitancy; peer mentor; community advisory board
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to intervention or control group; repeated measure assessments at 0 weeks, 14 weeks, and 18 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): non-intervention control (participants complete surveys only)
- Intervention (Experimental): Participants engage in weekly community-led small group discussions about health-related topics and answer surveys at 0, 14, and 18 week time points
  Interventions: Behavioral: Community-led discussion

INTERVENTIONS:
Behavioral: Community-led discussion — Participants engage in weekly community-led small group discussions about health related topics
  Arms: Intervention

SUMMARY:
The goal of this adapted intervention study is to assess how community-led group discussions about health-related topics may alter beliefs and intentions regarding healthcare recommendations, such as COVID-19 testing and vaccination.

DETAILED DESCRIPTION:
Eligible participants will be randomized to intervention or control group. Intervention group participants will meet virtually with other community member participants in small discussion groups once a week for 75 minutes over the course of 14 weeks. The online discussion groups will be led by peer mentor facilitators and supported by a research team member. Discussion topics will include current events and other health related topics. Control group participants will not meet in weekly discussion groups. At approximately the 0 weeks, 14 weeks, and 18 weeks time points, all participants will answer online surveys about health related topics. At the 14 weeks and 18 weeks time points, all participants will also be asked to self-administer a COVID-19 test that investigators provide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Resident of one of the 9 housing authority agencies
* Willing to participate in Zoom meetings and complete online assessments at baseline, 14-week, and 18-week timepoints
* Ability to read, speak, and understand English

Exclusion Criteria:

* May not have participated in Study 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Openness to COVID-19 Testing | 0 weeks, 14 weeks, 18 weeks
  The COVID-19 Testing Openness Questionnaire is an 7-item self-report measure designed to assess participants' openness to getting tested for COVID-19. Each item is rated on a 5-point scale, from 1 "Strongly Disagree" to 5 "Strongly Agree," with the sum of scores ranging from 7 to 35. Higher scores indicate greater openness to COVID-19 testing.
COVID-19 Testing Efficacy | 0 weeks, 14 weeks, 18 weeks
  The COVID-19 Testing Efficacy Scale is a 6-item self-report measure that will assess participants' perceived self- and response-efficacy related to COVID-19 testing. Each item is rated on a 5-point scale ranging from 1 "Strongly Disagree" to 5 "Strongly Agree," with the sum of scores ranging between 6 and 30. Higher scores indicate greater efficacy.
COVID-19 Trust | 0 weeks, 14 weeks, 18 weeks
  The COVID-19 Trust Questionnaire is an 18-item self-report measure to assess participants' trust of information provided by various institutions and individuals relating to COVID-19. Each item is rated on a 5-point Likert scale, with the sum of scores ranging from 18 to 90. Higher scores indicate greater trust.

SECONDARY OUTCOMES:
COVID-19 Vaccine Hesitancy | 0 weeks, 14 weeks, 18 weeks
  The Vaccine Hesitancy Questionnaire (VHQ) is an 18-item self-report measure that will assess participants' COVID-19 vaccine hesitancy. The VHQ was adapted from the Parent Attitudes about Childhood Vaccines (PACV) survey and contains 4 subscales: Immunization Behavior, Beliefs about Vaccine Safety and Efficacy, Attitudes about Vaccine Mandates and Exemptions, and Trust. Scores range from 11 to 85, with higher scores indicating greater hesitancy.
Social Connectedness | 0 weeks, 14 weeks, 18 weeks
  The Social Connectedness Scale Revised is a 20-item scale that measures a participant's feeling of connection with other people and their community. Each item is rated on a 6-point scale ranging from 1 "Strongly Disagree" to 6 "Strongly Agree," with the sum of scores ranging between 20 and 120. Higher scores indicate greater connectedness.
Health Literacy | 0 weeks, 14 weeks, 18 weeks
  The Health Literacy Scale (HLS-14) for Adults is a 14-item scale adapted for use in the US that measures an individual's ability to understand, access, and apply health-related information. Each item is rated on a 5-point scale ranging from 1 "Strongly Disagree" to 5 "Strongly Agree," with the sum of scores ranging between 14 and 70. Higher scores indicate greater health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli J England, PhD, Principal Investigator — Old Dominion University
Locations (1):
- Macon & Joan Brock Virginia Health Institute at Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No